CLINICAL TRIAL: NCT03182062
Title: Postoperative Complication and Hospital Stay Reduction With a Individualized Perioperative Lung Protective Ventilation During One-lung Ventilation: A Prospective, Multicenter, Randomized Trial
Brief Title: Individualized Perioperative Open-Lung Ventilatory Strategy During One-Lung Ventilation
Acronym: iPROVE-OLV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, Principal Investigador, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: iPROVE-OLV
Record Dates: First submitted 2017-05-25; First posted 2017-06-09 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Thoraric Surgery; Surgery Time Expected More Than Two Hours
Keywords: one lung ventilation; postoperative pulmonary complication; perioperative lung protective ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OLA-iHFNC (Active Comparator): Intraoperatively ventilated patients with a tidal volume (VT) of 5-6ml / kg of ideal body weight and respiratory rate to maintain normal carbon dioxide. After intubation, in all patients will be performed an alveolar recruitment maneuver (MRA) and a PEEP titration trial (see Calculation of optimal PEEP). Every 40 minutes will be assessed the need to adjust the level of PEEP by evaluating the dynamic compliance of the respiratory system (Crs). Faced with a decline in Crs> 10% a new MRA and optimal PEEP setting will be assessed.
  Postoperatively, high flow oxygen therapy will be individually indicated by evaluating peripheral oxygen saturation.
  Interventions: Procedure: Alveolar recruitment maneuver; Procedure: PEEP Titration Trial
- STD-O2 (Active Comparator): Intraoperatively ventilated patients with a tidal volume of 5-6 ml / kg of ideal body weightand respiratory rate to maintain normal carbon dioxide, PEEP 5 cmH2O. In this group no recruitment maneuvers or optimal PEEP setting will be performed.
  Postoperatively, standard oxygen therapy.
  Interventions: Procedure: Lung protective ventilation

INTERVENTIONS:
Procedure: Alveolar recruitment maneuver — To start the Alveolar Recruitment Maneuver (ARM) the ventilatory mode will be changed to pressure-controlled mode (PCV) with 20 cmH2O pressure control ventilation. A respiratory rate (RR) of 15 rpm, inspiration: expiration ratio of 1:1, FiO2 of 0.8 and PEEP of 5 cmH2O. The PEEP level will be increased in 5 cmH2O steps every 10 respiratory cycles, increasing to 15 cycles in the last level of PEEP (20 cmH2O), getting an opening pressure at 40 cmH2O airway (duration of the maneuver: 160 sec.)
  Arms: OLA-iHFNC
Procedure: PEEP Titration Trial — The ventilation mode will then switch back to volume controlled ventilation with the same baseline settings but with 20 cmH2O PEEP level. Then PEEP will be reduced in 2 cmH2O steps each maintained for 5 breaths the level of PEEP with the best (higher) dynamic compliance.
  Arms: OLA-iHFNC
Procedure: Lung protective ventilation — Ventilatory strategy with a PEEP level of 5 cmH2O but without recruitment maneuvers and PEEP titration trial.
  Arms: STD-O2

SUMMARY:
The purpose of this study is to determine whether individualized ventilatory management during one-lung ventilation in patients scheduled for thoracic surgery, combining the use of low tidal volumes, alveolar recruitment maneuvers, individually titrated positive end-expiratory pressure and individually indicated ventilatory support will decrease postoperative pulmonary complications, ICU and hospital length of stay compared to a standardized Lung Protective Ventilation (LPV).

ELIGIBILITY:
Inclusion Criteria:

* Planned thoracic surgery > 2 hours.
* Signed informed consent for participation in the study.

Exclusion Criteria:

* Age less than 18 years.
* Pregnant or breast-feeding.
* Patients with BMI >35.
* Syndrome of moderate or severe respiratory distress: PaO2/FiO2 < 200 mmHg.
* Heart failure: NYHA IV.
* Hemodynamic failure: CI <2.5 L/min/m2 and / or requirements before surgery ionotropic support.
* Diagnosis or suspicion of intracranial hypertension (intracranial pressure> 15 mmHg).
* Mechanical ventilation in the last 15 days.
* Presence of pneumothorax. Presence of giant bullae on chest radiography or computed tomography (CT).
* Patient with preoperatively CPAP.
* Participation in another experimental protocol at the time of intervention selection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2018-09-08 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Reduction of postoperative pulmonary complications | Up to 7 postoperative days
  composite of pulmonary infection, severe respiratory failure, acute respiratory distress syndrome, pneumothorax, bronchopleural fistula, atelectasis requiring bronchoscopy, empyema.

SECONDARY OUTCOMES:
Reduction of composite of postoperative pulmonary complications | Up to 30 postoperative days
  suspicion of pulmonary infection, mild acute respiratory failure, severe respiratory failure, acute respiratory distress syndrome
Reduction of composite of postoperative complications | Up to 7 and 30 postoperative days
  Renal failure, cardiac failure, sepsis, septic shock, surgical site infection, urinary infection and other pulmonary complications not included in the primary outcome such as leaks, atelectasis, pleural effusion, empyema, dyspnea.
Intensive care unit and hospital length of stay reduction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Javier Belda, MD, PhD, Study Director — Department of Anesthesia and Critical Care; Hospital Clinico Universitario
Locations (4):
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Gregorio Marañón, Madrid
  - Hospital clínico universitario, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ferrando C, Mugarra A, Gutierrez A, Carbonell JA, Garcia M, Soro M, Tusman G, Belda FJ. Setting individualized positive end-expiratory pressure level with a positive end-expiratory pressure decrement trial after a recruitment maneuver improves oxygenation and lung mechanics during one-lung ventilation. Anesth Analg. 2014 Mar;118(3):657-65. doi: 10.1213/ANE.0000000000000105. PMID 24557111
- [Result] Fleisher LA, Linde-Zwirble WT. Incidence, outcome, and attributable resource use associated with pulmonary and cardiac complications after major small and large bowel procedures. Perioper Med (Lond). 2014 Oct 7;3:7. doi: 10.1186/2047-0525-3-7. eCollection 2014. PMID 25313335
- [Result] Licker MJ, Widikker I, Robert J, Frey JG, Spiliopoulos A, Ellenberger C, Schweizer A, Tschopp JM. Operative mortality and respiratory complications after lung resection for cancer: impact of chronic obstructive pulmonary disease and time trends. Ann Thorac Surg. 2006 May;81(5):1830-7. doi: 10.1016/j.athoracsur.2005.11.048. PMID 16631680
- [Derived] Zorrilla-Vaca A, Barbeta E, Librero J, Ferrando C; iPROVE-OLV Research Network Group. Open-lung ventilation and mechanical power in thoracic surgery: Post hoc analysis of a multicentre randomised trial. Eur J Anaesthesiol. 2025 Sep 4. doi: 10.1097/EJA.0000000000002271. Online ahead of print. PMID 40905246
- [Derived] Mazzinari G, Diaz-Cambronero O, Garutti I, Errando CL, Ferrando C; iPROVE-OLV investigators. Impact of neuromuscular block monitoring and reversal on postoperative pulmonary complications in thoracic surgery: a Bayesian analysis of the iPROVE-OLV trial. Br J Anaesth. 2025 Nov;135(5):1428-1440. doi: 10.1016/j.bja.2024.11.041. Epub 2025 Feb 1. PMID 39893063
- [Derived] Ferrando C, Carraminana A, Pineiro P, Mirabella L, Spadaro S, Librero J, Ramasco F, Scaramuzzo G, Cervantes O, Garutti I, Parera A, Argilaga M, Herranz G, Unzueta C, Vives M, Regi K, Costa-Reverte M, Sonsoles Leal M, Nieves-Alonso J, Garcia E, Rodriguez-Perez A, Farina R, Cabrera S, Guerra E, Gallego-Ligorit L, Herrero-Izquierdo A, Valles-Torres J, Ramos S, Lopez-Herrera D, De La Matta M, Gokhan S, Kucur E, Mugarra A, Soro M, Garcia L, Sastre JA, Aguirre P, Salazar CJ, Ramos MC, Morocho DR, Trespalacios R, Ezequiel-Fernandez F, Lamanna A, Pia Cantatore L, Laforgia D, Bellas S, Lopez C, Navarro-Ripoll R, Martinez S, Vallverdu J, Jacas A, Yepes-Temino MJ, Belda FJ, Tusman G, Suarez-Sipmann F, Villar J; iPROVE-OLV Research Network Group. Individualised, perioperative open-lung ventilation strategy during one-lung ventilation (iPROVE-OLV): a multicentre, randomised, controlled clinical trial. Lancet Respir Med. 2024 Mar;12(3):195-206. doi: 10.1016/S2213-2600(23)00346-6. Epub 2023 Dec 5. PMID 38065200